CLINICAL TRIAL: NCT02776228
Title: The Influence of Short Term Treatment With Benzodiazepine After Cardiac Surgery
Brief Title: Treatment With Benzodiazepine After Cardiac Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: cs 001-16
Record Dates: First submitted 2016-03-23; First posted 2016-05-18 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-11

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — brotizolam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- benzodiazepine (Experimental): The patient which will be in the Experimental arm (after randomization) will receive 0.25 mg of Brotizolam (short acting benzodiazepine) for six weeks from the day of discharge.
  Interventions: Drug: Brotizolam
- placebo (Placebo Comparator): The patient which will be in the placebo arm (after randomization) will receive placebo for six weeks from the day of discharge.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Brotizolam — Every patient which will enroll to the study will fill up The Pittsburgh Sleep Quality Index in there admission to the cardiac surgery unit. in the discharge day the patient will receive 0.25 mg brotizolam once a day before sleep for six weeks. one week and six weeks after discharge day, there is routine follow up in our outpatient clinic. in those appointed time the patient will fill again The Pittsburgh Sleep Quality Index.
  Other Names: Lendormin
  Arms: benzodiazepine
Drug: placebo — Every patient which will enroll to the study will fill up The Pittsburgh Sleep Quality Index in there admission to the cardiac surgery unit. in the discharge day the patient will receive 0.25 mg LACTOSE once a day before sleep for six weeks. one week and six weeks after discharge day, there is routine follow up in our outpatient clinic. in those appointed time the patient will fill again The Pittsburgh Sleep Quality Index.
  Arms: placebo

SUMMARY:
The study deals with the prevalence of insomnia after heart surgery and the outcome of treatment with Benzodiazepine for this phenomena.

DETAILED DESCRIPTION:
Patients after heart surgery develop sleep disorder in the form of Insomnia. This finding is known and described in the literature with respect to a large number of major operations such as the pneumonectomy, esophageal resection, pancreatic surgery, liver surgery and so on. In the general population, Insomnia is a common disorder and describe in more than 50% in adults over the age of 50. In patients with comorbidity among other things, heart disease indicates a rate of up to 85% of chronic insomnia. The reasons for insomnia after multiple heart surgery, including emotional stress that accompanies the patient after surgery, pain and prolonged hospitalization in the hospital. In this study, aim to compare the results of short-term treatment with sleep medication after heart surgery on morbidity and immediate recovery. This study will allow us to examine the effect of sleep medication therapy in patients receiving treatment compared to patients who did not receive treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and older.
2. Applicants hospital for open heart surgery

Exclusion Criteria:

1. patients who came to emergency heart surgery.
2. patients who are not hemodynamically or respiratory stable
3. Patients who were taking hypnotic drugs on a daily basis before surgery.
4. Patients with low compliance that will not be able to fill out a sleep diary
5. lactose intolerance (due to components placebo)
6. Patients who can not take medication by one or more of the following:

   * pregnant.
   * nursing.
   * Patients with severe respiratory insufficiency
   * Patients with liver failure.
   * Patients who are addicted to alcohol
   * Patients without psychiatric background.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Assessing chronic insomnia | 1 year
  The following outcome will be evaluated by Pittsburgh sleep quality index questionnaire before heart surgery.

SECONDARY OUTCOMES:
Reducing insomnia in post cardiac surgery | 1 year
  The following outcome will be evaluated by Pittsburgh sleep quality index questionnaire after heart surgery.

CONTACTS AND LOCATIONS:
Overall Officials: gil mr bolotin, MD, Principal Investigator — Rambam Health Care Campus

IPD SHARING:
Plan to Share IPD: Yes